CLINICAL TRIAL: NCT00674934
Title: Phase 1 Study to Determine the Efficacy of Using Far Infrared Radiation for Multiple Sclerosis.
Brief Title: Far Infrared Irradiation for Managing and Treating Multiple Sclerosis (MS)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GAAD Medical Research Institute Inc. (Other)
Responsible Party: Dr. Kwasi Donyina/Founder & President, GAAD Medical Research Institute Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAAD-MS-CTP1
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Last update posted 2009-01-05 (Estimated); Status verified 2009-01

CONDITIONS: Multiple Sclerosis
Keywords: MS (Multiple Sclerosis); Multiple Sclerosis, Acute Fulminating; Sclerosis, Disseminated
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Radiation
  Interventions: Radiation: Far Infrared Radiation (5μm to 20μm wavelength)

INTERVENTIONS:
Radiation: Far Infrared Radiation (5μm to 20μm wavelength) — Far Infrared Radiation (5μm to 20μm wavelength). Far Infrared radiation for 30 to 40 minutes per treatment session.
  Other Names: Far Infrared Radiation

SUMMARY:
Multiple sclerosis (abbreviated MS) is an autoimmune condition in which the immune system attacks the central nervous system (CNS), leading to demyelination. This study will investigate the use of far infrared radiation for MS control, management and treatment.

DETAILED DESCRIPTION:
MS a demyelinating disease, is any disease of the nervous system in which the myelin sheath of neurons is damaged. This impairs the conduction of signals in the affected nerves, causing impairment in sensation, movement, cognition, or other functions depending on which nerves are involved.

MS affects the areas of the brain and spinal cord known as the white matter. White matter cells carry signals between the grey matter areas, where the processing is done, and the rest of the body. More specifically, MS destroys oligodendrocytes which are the cells responsible for creating and maintaining a fatty layer, known as the myelin sheath, which helps the neurons carry electrical signals.

Observations from our research studies indicate that, far infrared rays provide energy to the body, improve the autonomic functions of the nervous system, restore the functions of the endocrine system, strengthen the immune system, improve blood circulation and increase the level of oxygen in the cells and promote the regeneration of muscle cells, nerves and brain cells.

It is hereby postulated that irradiation using far infrared, with wavelength between 5 to 20 microns, of the central nervous system, the endocrine system and the whole body could prevent, control, manage or possibly lead to complete rehabilitation of people who have MS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MS

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-05 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Treatment of MS | 2 years

SECONDARY OUTCOMES:
Rehabilitation of MS Patients | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Ken Nedd, M.D., Principal Investigator — GAAD Medical Research Institute Inc.
Locations (1):
- The Centre for Incurable Diseases, Toronto, Ontario, Canada